CLINICAL TRIAL: NCT02411253
Title: European Phase-IIb Clinical Trial Evaluating Efficacy of Low Dose rhIL-2 in Patients With Recently-diagnosed Type 1 Diabetes DIABIL-2
Brief Title: Low-dose rhIL-2 in Patients With Recently-diagnosed Type 1 Diabetes
Acronym: DIABIL-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Iltoo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P121001
Record Dates: First submitted 2015-03-23; First posted 2015-04-08 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Type 1 Diabetes
Keywords: IL2; Interleukin 2; IL-2; Auto-immune disease; Insulin; Diabetes; Regulatory T cells; Treg; Immunoregulation; Immune tolerance; Immunotherapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhIL-2 (Experimental): * 0.5 MIU/m²/day of IL2 with a maximum of 1MIU/day in a volume of 1 ml for children and adolescents,
  * 1MIU/day for adults.
  Subcutaneous injection every day (5 days) then:
  * Regimen A injection every two weeks between D15 and D351,
  * Regimen B injections every week between D15 and D351
  Interventions: Drug: rhIL-2
- Placebo (Placebo Comparator): Placebo with a identical formulation and regimen of injections i.e. Subcutaneous injection every day (5 days) then:
  * Regimen A injection every two weeks between D15 and D351
  * Regimen B injections every week between D15 and D351
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: rhIL-2 — Subcutaneous injections of IL2 according to regimen A Subcutaneous injections of IL2 according to regimen B
  Arms: rhIL-2
Drug: Placebo — Subcutaneous injections of Placebo according to regimen A Subcutaneous injections of Placebo according to regimen B
  Arms: Placebo

SUMMARY:
Type 1diabetes (T1D) is caused by autoimmune destruction of the pancreatic islet ß-cells, leading to an absolute deficiency in insulin.

In health, regulatory T cells (Tregs) suppress immune responses against normal tissues, and likewise prevent autoimmune diseases. Tregs are insufficient in T1D.

The investigators previously showed that administration of low doses of IL-2 induces selective expansion and activation of Tregs in mice and humans.

The investigators hypothesize that Tregs expansion and activation with low doses of IL2 could block the ongoing autoimmune destruction of insulin producing cells in patients with recently diagnosed T1D.

DETAILED DESCRIPTION:
Scientific justification:

Clinical and preclinical studies, together with supportive mechanistic data showing that Tregs are activated by much lower IL-2 concentration than effector T cells (Teffs), provide a strong rationale for studying efficacy of low dose IL2 to stop the autoimmune destruction of insulin-secreting beta cells in patient with recently diagnosed with T1D.

Primary objective:

1. To evaluate efficacy of low dose IL-2 for the preservation of residual pancreatic β cells function
2. To select the optimal regimen of administration of IL-2

Primary assessment criterion:

AUC (T0-T120) of serum C-peptide, determined after a mixed meal tolerance test at month 12, compared to baseline.

Secondary objectives:

1. To assess Tregs expansion after an induction period and during maintenance therapy
2. To assess safety of IL-2 during the treatment period (1 year) and 1 year after its discontinuation
3. To assess the relation between Tregs expansion and preservation of residual pancreatic β cells function
4. To assess clinical and biological responses according to (i) pubertal stage group, (i) time from diagnosis to treatment initiation, (iii) biomarkers of responses
5. To assess effects of IL-2 on disease-specific immune responses
6. To identify biomarkers for predicting/monitoring safety and efficacy of IL-2.

Secondary assessment criteria:

* Serum concentrations of C-peptide
* AUC (T0-T120) of serum C-peptide after a mixed meal tolerance test after treatment discontinuation
* Diabetic monitoring (insulin use)
* HbA1c and IDAA1c score
* Number of hypoglycaemic episodes (< 0.5 g/L on capillary sample) over 15 days before each visit.
* Number of clinically significant symptomatic episodes of hypoglycaemia between each visit.
* Change in Tregs (expressed as percentage of CD4 and absolute numbers) at day 5 compared to baseline.
* Change in trough level of Tregs (%CD4+ and absolute numbers) at month 1, month 3, month 6, month 9, month 12, compared to baseline; and then month 15 and 24 after treatment discontinuation.
* Change in Foxp3 gene methylation
* Cytokines and chemokines assays at day 5, month 1, month 3, month 6, month 9, and month 12 compared to baseline and then month 15 and month 24 after treatment discontinuation.
* Transcriptome analysis.
* Genotyping at baseline
* Treg phenotype and functionality in adults and adolescents only including pStat5 analysis

Pharmacokinetic of IL2 will be performed (in patients from regimen A only) on day 1 at T0, T60min (1h), T120min (2h), T240min (4h), T360min (6h), T600min (10h), T1440min (24h=day2) on day 4, V8 (D29±1day) and V54 (day 351±3 days) at the same time points in 27 patients of regimen A.

• Safety parameters will be evaluated by clinical examination (including height/weight and pubertal stage especially for children and adolescents), routine laboratory tests, ILT-101 auto-antibodies, ancillary investigations and adverse event.

Experimental design:

This is a multicenter European, sequential-group, randomized, double-blind trial evaluating IL-2 versus placebo

Population involved:

Male or female, aged between 6 and 35 years, with type 1 diabetes diagnosed for less than two months.

Number of subjects: 138

Inclusion period: 49 months

Duration of patient participation: 24 months (treatment period: 12 months, follow-up period: 12months)

Total duration of the study: 73 months

Statistical analysis:

The principal efficacy analysis will be drawn from the intention to treat group.

The per-protocol analysis will be used to confirm the intention to treat analysis.

For each regimen:

- MMTT: C-peptide concentrations will be summarized by the AUC from T0 to T+120 min. Before statistical analysis, log (x+1) normalizing transformation will be used, and IL-2 and placebo treated patients will be compared using a mixed model of ANCOVA including baseline value as covariate and factor pubertal stage group.

Quantitative endpoints will be analyzed using same methods as primary endpoint. Categorical endpoints will be analyzed using multivariate logistic regression models.

Subgroups analyses: Response to treatment will be analysed according to criteria such as:

* Pubertal stage, age, gender, BMI…
* Biomarkers (identified in previous studies as predictive of patients' response to treatment)

Funding source: European Commission under the Health Cooperation Programme of the Seventh Framework Programme (Grant Agreement n°305380-2).

ELIGIBILITY:
Inclusion criteria

* Age 6-35 years old.
* Male or female both using effective methods of contraception during treatment if sexually active.
* Specifically; Females (if sexually active) with childbearing potential must use contraceptive methods that are considered as highly-effective (pearl index < 1). The following methods are acceptable: Oral , injectable, or implanted hormonal contraceptives (with the exception of oral minipills ie low-dose gestagens which are not acceptable (lynestrenol and norestisteron), Intrauterine device, Intrauterine system (for example, progestin-releasing toit),
* beta HCG negative at inclusion;
* With type-1 diabetes:
* Newly diagnosed (ADA criteria, see annexe 19.6) at most three months between insulin initiation and anticipated start of experimental treatment.
* Positive for one or more of the autoantibodies typically associated with T1D (anti-islet, -insulin, -GAD, -IA2, -ZnT8)
* With a detectable peak C-peptide concentration during a standardised MMTT at Visit MMTT (≥0.2pmol/ml);
* patients with a stable blood glucose level and seric glycaemia between 60 mg/dL and 250 mg/dL verified at MMTT visit
* Absence of clinically significant abnormal laboratory values (out of range and associated with clinical symptoms or signs) in haematology, biochemistry, thyroid, liver and kidney function;
* Normal cardiac function: no documented history of heart disease and absence of family history of sudden death, normal ECG especially QTc duration within normal value (<480ms);
* Free, informed and written consent, signed by the patient and investigator before any Study examination. If the patient is a minor by child and both parents or child and the legal representative in case only one parent is alive. (Journal officiel des communautés européennes (1.5.2001)
* NB: patient with history of thyroidism on treatment at the inclusion and with normal thyroid hormone values (TSH+T4) can be included.

Exclusion criteria

* Children under the age of 6 years old cannot be included
* Patient who, before inclusion, have been treated with other anti-diabetic medication than Insulin for more than 3 months consecutively
* Chronic adrenal insufficiency known or fasting ACTH ≥2.5 ULN normal at inclusion after control;
* Anti TPO present at inclusion and abnormal TSH and T4
* Anti-transglutaminase positive at inclusion
* Hypersensitivity to the active substance or to any of the excipients
* Any major health problem including: any major auto-immune/auto-inflammatory disease (other than type 1 diabetes) present at inclusion, any significant respiratory disease (such as moderate or severe COPD or asthma) requiring the chronic use of corticosteroids (whatever route of administration) and serious digestive malfunctions.
* Patient with existing malignancy or history of malignancy
* Major psychosocial instability with expected lack of compliance with insulin treatment, psychiatric pathology of patient or parents, or major problems of family dynamics;
* Signs of active infection;
* Any patient with obesity defined as BMI ≥ 35
* Existence of a serious malfunction of a vital organ;
* History of organ allograft;
* Use of treatments not allowed in the Study (see Section 8.4.2);
* Vaccination with alive attenuated virus within 4 weeks of the first injection of the induction period and during the whole maintenance period
* Pregnant female (confirmed by laboratory testing) or lactating
* Participation in another clinical trial in the previous 3 months;
* Lack of affiliation to a social security scheme (as a beneficiary or assignee).

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
AUC (T0-T120) of serum C-peptide, determined after a mixed meal tolerance test at month 12, compared to baseline. | Baseline, month12

SECONDARY OUTCOMES:
Serum concentrations of C-peptide | month 3, month 6, month 9, month 15
AUC (T0-T120) of serum C-peptide after a mixed meal tolerance test after treatment discontinuation | month 15
Diabetic monitoring (insulin use) | baseline, Day 1, Day 5, month 1, month 3, month 6, month 9, month 12, month 15, month 18, month 21.
HbA1c and IDAA1c score | baseline, month 3, month 6, month 9, month 12, month 15
Number of hypoglycaemic episodes (< 0.5 g/L on capillary sample) over 15 days before each visit. | baseline, Day 1, Day 5, month 1, month 3, month 6, month 9, month 12, month 15, month 18, month 21
Number of clinically significant symptomatic episodes of hypoglycaemia between each visit. | baseline, Day 1, Day 5, month 1, month 3, month 6, month 9, month 12, month 15, month 18, month 21
Change in Tregs (expressed as percentage of CD4 and absolute numbers) at day 5 compared to baseline. | Baseline, Day 5.
Change in trough level of Tregs (%CD4+ and absolute numbers) at month 1, month 3, month 6, month 9, month 12, compared to baseline; and then month 15 and 24 after treatment discontinuation. | Baseline, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, Month 24
Change in Foxp3 gene methylation | Day 1, Day 5, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15
Cytokines and chemokines assays at day 5, month 1, month 3, month 6, month 9, and month 12 compared to baseline and then month 15 and month 24 after treatment discontinuation. | Baseline, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, Month 24
Transcriptome analysis. | Baseline, Month 6, Month 12
  Transcriptome analysis on whole PBMCs will allow analysis of changes in inflammation-related signatures, as already described in Saadoun et al. NEJM, 2011.
Genotyping at baseline | baseline
  Genotyping will be used to assess genetic variation (polymorphisms) associated with T1D, such as those linked to IL2RA, PTPN22, CTLA-4...
Treg phenotype and functionality in adults and adolescents only including pStat5 analysis | Day 1, Day 5, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15
Clinical examination. | Baseline Day 1, Day 5, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Height/weight and pubertal stage especially for children and adolescents. | Baseline, Month 12, Month 24
  Based on Tanner staging (Tanner J. M. 1986).
Routine laboratory tests | Baseline Day 1, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
  Biochemistry, Liver function
Haematology | Baseline Day 1, Day 5, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Detection of IL-2 auto-antibodies | Day1, Month 6, Month 12
T cells repertory | Day 1, Day 5, Month 6, Month 12
Intestinal microbiota. | Baseline, Month 6, Month 12
Adverse event. | Baseline, Day 1, 2, 3, 4, 5, Month 1, Month 3, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
  Throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: David Klatzmann, MD, Ph.D., Study Director — Assistance Publique - Hôpitaux de Paris
Locations (34):
- Belgium (3):
  - Pediatric Department, Centre Hospitalier Régional de la Citadelle, Liège, Province De Liège
  - UZ - Diabetes voor Kinderen en Adolescenten-Leuven, Leuven
  - CHU UCL Namur - site Godinne, Yvoir
- France (25):
  - Centre d'Investigations Cliniques, CHU-HOPITAL HAUTEPIERRE, Strasbourg, Alsace
  - Centre d'Investigations Cliniques, HÔPITAL CIVIL, Strasbourg, Alsace
  - Service de pédiatrie 1CHU de HAUTEPIERRE, Strasbourg, Alsace
  - Structure d'Endocrinologie-Diabète-Nutrition et Addictologie HOPITAUX UNIVERSITAIRES NHC, Strasbourg, Alsace
  - Service d'endocrinologie, diabétologie, maladies métaboliques, et nutrition, CHU de Bordeaux, Hôpital Haut Levêque, Pessac, Aquitaine
  - Service d' Endocrinologie HOPITAL CAVALE BLANCHE, Brest, Brittany Region
  - Service de Pédiatrie, HOPITAL MORVAN, Brest, Brittany Region
  - Service de Pédiatrie CHRU DE NANTES, Nantes, Brittany Region
  - Service d' Endocrinologie Diabétologie CHRU DE RENNES, Rennes, Brittany Region
  - Médecine pédiatrique, CHU Jean Minjoz, Besançon, Franche-Compté
  - Service Diabétologie -Endocrinologie, CHU Jean Minjoz, Besançon, Franche-Comté
  - CHRU de Lille, Hôpital Claude Huriez Service d'endocrinologie, Lille, Hauts-de-France
  - Service Pédiatrie - Gastro-entérologie, Hépatologie, Nutrition, Diabétologie, Hôpital des Enfants Pôle Enfants, Toulouse, Midi Pyrénnées
  - Service d' Endocrinologie, maladies métaboliques HOPITAL NORD, Marseille, PACA
  - Service de Nutrition - Maladies Métaboliques - Endocrinologie HOPITAL DE LA CONCEPTION, Marseille, PACA
  - Hopital G&R Laënnec , Endocrinologie, Maladies Métaboliques et Nutrition, Saint-Herblain, Pays de la Loire Region
  - Unité d'Endocrinologie et Diabétologie Pédiatriques, CHU de Marseille, Hôpital La Timone Enfants, Marseille, Provence-Alpes-Côte d'Azur Region
  - Endocrinologie-Diabétologie-Maladies de la nutrition, Centre Hospitalier Lyon-Sud, Lyon, Rhones-Alpes
  - Service d'Endocrinologie pédiatrique - HFME, Bron
  - CIC Paris-Est (Adultes), Hôpitaux Universitaires Pitié-Salpêtrière, Charles Foix, Paris, Île-de-France Region
  - Institut E3M, Hôpital Pitié-Salpêtrière, Paris, Île-de-France Region
  - CIC pédiatrique Hôpital Necker Enfants Malades, Paris, Île-de-France Region
  - Endocrinologie gynécologie diabétologie pédiatriques, Hôpital Universitaire Necker Enfants Malades., Paris, Île-de-France Region
  - CIC Pédiatrique, Hôpital d'enfants Robert Debré, Paris, Île-de-France Region
  - Service d'Endocrinologie Pédiatrique, Hôpital d'enfants Robert Debré, Paris, Île-de-France Region
- Germany (3):
  - Division of Endocrinology and Diabetology, Department of Internal Medicine II, University Hospital of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Division of Endocrinology, Diabetology and Metabolic Diseases, University Hospital of Freiburg, Department for children and adolescents, Freiburg im Breisgau, Baden-Wurttemberg
  - Institute of Diabetes Research, Helmholtz Zentrum München, München, Bavaria
- Center for Pediatric and Adolescent Diabetes Care and Research, Rotterdam, Randstad Holland, Netherlands
- Dept. of Clinical Sciences Lund University, Skåne University Hospital., Malmo, Öresund Region, Sweden
- Endocrinology and Diabetes department, University Hospital of Basel, Basel, Canton of Basel-City, Switzerland